CLINICAL TRIAL: NCT00385112
Title: Follow Up on Freestyle Valves for Right Ventricular Outflow Tract Reconstruction in Children
Brief Title: Follow Up on Freestyle Valves in Children
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kirk R. Kanter, MD, Chief, Pediatric Cardiac Surgery, Emory University
Other Study IDs: IRB00000124; 06-138
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Right Ventricle; Pulmonary Valve Stenosis; Pulmonary Valve Atresia
Keywords: Cardiology; Echocardiograms; Surgery; Valve Disease; Heart Valve Disease
MeSH Terms: conditions — Pulmonary Valve Stenosis; Pulmonary Atresia; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Echocardiogram — 2D echocardiogram with Doppler flow

SUMMARY:
The purpose of this study is to determine if the Medtronic Freestyle porcine valve is effective over a long period of time when it is used to replace the valve that normally allows blood to flow from the right lower pumping chamber of the heart to the lungs.

DETAILED DESCRIPTION:
During the time between June 1998 and June 2006, the Medtronic Freestyle® porcine aortic root (Medtronic, Minneapolis, MN) was used for reconstruction of the right ventricular outflow tract in children that underwent surgery at Children's Healthcare of Atlanta. These children were born with heart problems that made it difficult for blood to flow from the lower right chamber of the heart to the lungs where it would normally pick up oxygen to be used by the body. Consequently, these children required surgery to repair the valve and eliminate this restriction of blood flow to the lungs in order to preserve life. In this case, the Freestyle valve was used. It is a relatively new valve and it is not known how it functions and how it impacts overall heart function over a long period of time. We are requesting permission to recruit volunteers that have received the Freestyle valve for this purpose in order to determine its long term performance. Specifically, we are seeking volunteers that are willing to have an echocardiogram performed. It is through the evaluation of a recent echocardiogram, as it compares to previous echocardiograms performed on the same patient, that the usefulness of the Freestyle valve will be evaluated for its durability and its long term impact on heart function.

ELIGIBILITY:
Inclusion Criteria

* Patients that have received the Medtronic Freestyle® porcine aortic root for right ventricular outflow tract reconstruction that have not had a standard of care echocardiogram performed in the last 12 months.
* Patients that have received the Medtronic Freestyle® porcine aortic root for right ventricular outflow tract reconstruction whose most recent echocardiogram is not useful for evaluating the study points despite the fact that it may have been performed within the last 12 months.
* Informed consent obtained from the legal guardian or patient if > 18 years of age.

Exclusion Criteria

* Patients that have not received the Medtronic Freestyle® porcine aortic root for right ventricular outflow tract reconstruction.
* Patients that are eligible to participate based on the previous criteria for whom informed consent is not obtained from the patient or legal guardian.

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients that have received the Medtronic Freestyle® porcine aortic root for right ventricular outflow tract reconstruction that have not had a standard of care echocardiogram performed in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2006-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
We hypothesize that this Medtronic Freestyle® porcine aortic root valve has good long term hemodynamic performance and longevity. | Retrospective Chart Review
  Retrospective Chart Review

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Kanter, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Result] Kanter KR, Fyfe DA, Mahle WT, Forbess JM, Kirshbom PM. Results with the freestyle porcine aortic root for right ventricular outflow tract reconstruction in children. Ann Thorac Surg. 2003 Dec;76(6):1889-94; discussion 1894-5. doi: 10.1016/s0003-4975(03)01304-3. PMID 14667606